CLINICAL TRIAL: NCT02951728
Title: Phase I/II Trial of Decitabine + R-CHOP in Diffuse Large B-Cell Lymphoma
Brief Title: Decitabine Plus R-CHOP in Diffuse Large B-cell Lymphoma
Acronym: DR-CHOP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DR-CHOP
Record Dates: First submitted 2016-10-24; First posted 2016-11-01 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Decitabine plus R-CHOP (Experimental): Rituximab 375 mg/m2 IV d6; Cyclophosphamide 750mg/m2 IV d7; Doxorubicin 50mg/m2 IV d7; Vincristine 1.4 mg/m2 IV d7; Prednisone 60 mg/m2 PO d7-11;
  Decitabine will be administered intravenously at dose levels as follow in Phase 1:
  Dose level 1: Decitabine 10 mg/m2 days 1-5; Dose level 2: Decitabine 15 mg/m2 days 1-5; Dose level 3: Decitabine 20 mg/m2 days 1-5 and determine the maximum tolerated dose.
  In phase 2, Decitabine will be administered intravenously at MTD.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Decitabine

INTERVENTIONS:
Drug: Rituximab
Drug: Cyclophosphamide
Drug: Doxorubicin
Drug: Vincristine
Drug: Prednisone
Drug: Decitabine

SUMMARY:
This is a Phase I/II Trial of Decitabine + R-CHOP in Diffuse Large B-Cell Lymphoma

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed DLBCL, CD20 positive.
* must have at least one site of measurable disease, 1.5 cm in diameter or greater.
* has not had any previous treatment.
* International Prognostic Index >1.
* Able to adhere to the study visit schedule and other protocol requirements.
* must have laboratory test results within these ranges: Absolute neutrophil count ≥1500/mm3 Platelet count≥75,000/mm3 Serum creatinine≤1.5×upper limit of normal (ULN) Total bilirubin≤1.5×ULN. Higher levels are acceptable if these can be attributed to active hemolysis or ineffective erythropoiesis.

AST (SGOT) and ALT (SGPT) ≤2×ULN

* Disease free of prior malignancies with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* Women of childbearing potential must have a negative serum pregnancy test prior to Decitabine treatment.
* Women of childbearing potential should be advised to avoid becoming pregnant and men should be advised to not father a child while receiving treatment with Decitabine. The effects of Decitabine on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Age 15 to 75 years.
* Ability to understand and the willingness to sign a written informed consent document.
* ECOG performance status of 0-2

Exclusion Criteria:

* Patients must not have any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Patients must not have any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Concurrent use of other anti-cancer agents or treatments.
* Known positive for HIV. If HbsAg positive, should check HBV DNA, DNA positive patients cannot be enrolled. If HBsAg negative but HBcAb positive (whatever HBsAb status), should check HBV DNA, DNA positive patients cannot be enrolled.
* Known central nervous system involvement by lymphoma.
* Known or suspected hypersensitivity to Decitabine or mannitol.
* Pregnant and lactating women are excluded from the study because the risks to an unborn fetus or potential risks in nursing infants are unknown.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-05 (Actual); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose | day1 to 21
  The primary endpoint for the phase I portion of the study is to determine the maximum tolerated dose of Decitabine when given in combination with a standard dose (q21 day) regimen of R-CHOP in patients with DLBCL.
complete response rate | 21 days after 6 cycles of treatment (each cycle is 21 days)
  The primary endpoint for the phase II portion of the study will be complete response rate.

SECONDARY OUTCOMES:
Overall response rate | 21 days after 6 cycles of treatment (each cycle is 21 days)
Event-free survival | 2 years
Overall survival | 2 years
Progression-free survival | 2 years
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Up to 30 days after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, MD，PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No